CLINICAL TRIAL: NCT04511702
Title: A Phase 4, Multicenter, Open-Label, Infusion Duration Study To Assess Safety, Tolerability and Efficacy of Pegloticase Administered With a Shorter Infusion Duration in Subjects With Uncontrolled Gout Receiving Methotrexate
Brief Title: Infusion Duration Study To Assess Tolerability of Pegloticase Administered With a Shorter Infusion Duration in Subjects With Uncontrolled Gout Receiving Methotrexate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-KRY-403
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Chronic Uncontrolled Gout; Gout; Uncontrolled Gout
Keywords: gout; uncontrolled gout
MeSH Terms: conditions — Gout | interventions — Pegloticase; Methotrexate

STUDY DESIGN:
Intervention Model Description: Three different infusion durations may be used. 60-minute infusion, 45-minute infusion and 30-minute.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pegloticase 60 Minute Infusion with methotrexate (MTX) (Experimental): Pegloticase 60 Minute Infusion with methotrexate (MTX). Participants will receive MTX (15 mg) (weekly) during the Run-in Period, then pegloticase (every 2 weeks) with MTX (weekly) for 24 weeks
  Interventions: Biological: Pegloticase with MTX
- Pegloticase 45 Minute Infusion with methotrexate (MTX) (Experimental): Pegloticase 45 Minute Infusion with methotrexate (MTX). Participants will receive MTX (15 mg) (weekly) during the Run-in Period, then pegloticase (every 2 weeks) with MTX (weekly) for 24 weeks
  Interventions: Biological: Pegloticase with MTX
- Pegloticase 30 Minute Infusion with methotrexate (MTX) (Experimental): Pegloticase 30 Minute Infusion with methotrexate (MTX). Participants will receive MTX (15 mg) (weekly) during the Run-in Period, then pegloticase (every 2 weeks) with MTX (weekly) for 24 weeks
  Interventions: Biological: Pegloticase with MTX

INTERVENTIONS:
Biological: Pegloticase with MTX — Participants will receive MTX during the run-in period then pegloticase with MTX for up to 24 weeks during the treatment period
  Other Names: Methotrexate

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficiency of pegloticase administered with a shorter infusion duration in participants with uncontrolled gout receiving methotrexate.

DETAILED DESCRIPTION:
Approximately 180 participants will be enrolled. After a 4-week methotrexate run-in period, participants will be treated for up to 24 weeks with weekly oral methotrexate and biweekly 8mg pegloticase infusions. Up to three pegloticase infusion durations will be assessed in the study: 60-minute infusion, 45-minute infusion and 30-minute infusion. Safety evaluations will be performed regularly throughout the course of the study.

Acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women ≥18 years of age.
2. Uncontrolled gout, defined as meeting the following criteria:

   * Hyperuricemia during the screening period defined as sUA ≥6 mg/dL
   * Failure to maintain normalization of sUA with xanthine oxidase inhibitors at the maximum medically appropriate dose, or with intolerable side effects or a contraindication to xanthine oxidase inhibitor therapy based on medical record review or subject interview.
   * Symptoms of gout including at least 1 of the following:

     * Presence of at least one tophus
     * Recurrent flares defined as 2 or more flares in the past 12 months prior to screening
     * Presence of chronic gouty arthritis
3. Willing to discontinue all oral urate-lowering therapy at least 7 days prior to MTX dosing at Week -4 and remain off of urate lowering therapy when receiving pegloticase infusions during the study.

Exclusion Criteria:

1. Severe chronic or recurrent bacterial infections, such as recurrent pneumonia or chronic bronchiectasis.
2. Current or chronic treatment with systemic immunosuppressive agents such as MTX, azathioprine, or mycophenolate mofetil; prednisone ≥10 mg/day or equivalent dose of other corticosteroid on a chronic basis (defined as 3 months or longer) would also meet exclusion criteria.
3. Glucose-6-phosphate dehydrogenase (G6PD) deficiency (tested at Screening Visit).
4. Severe chronic renal impairment (estimated glomerular filtration rate <40 mL/min/1.73 m2) at the Screening Visit based on 4 variable-Modification of Diet in Renal Disease [MDRD] formula or currently on dialysis.
5. Non-compensated congestive heart failure or hospitalization for congestive heart failure or treatment for acute coronary syndrome (myocardial infarction or unstable angina) within 3 months of the Screening Visit, or current uncontrolled arrhythmia, or current uncontrolled blood pressure (BP) (>160/100 mmHg) prior to Week -4.
6. Pregnant, planning to become pregnant, breastfeeding, planning to impregnate female partner, or not on an effective form of birth control, as determined by the Investigator.
7. Prior treatment with pegloticase (KRYSTEXXA), another recombinant uricase (rasburicase), or concomitant therapy with a polyethylene glycol-conjugated drug.
8. Currently receiving systemic or radiologic treatment for ongoing cancer.
9. History of malignancy within 5 years other than non-melanoma skin cancer or in situ carcinoma of cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (39):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Orthopedic Physicians Alaska, Anchorage, Alaska
  - Arizona Arthritis & Rheumatology Research, Gilbert, Arizona
  - Arthritis & Rheumatology Research, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, Phoenix, Arizona
  - Medvin Clinical Research, Covina, California
  - Amicis Research Center, Northridge, California
  - Providence Saint John's Health Center, Santa Monica, California
  - Medvin Clinical Research, Thousand Oaks, California
  - Medvin Clinical Research, Tujunga, California
  - University of Colorado Division of Rheumatology, Aurora, Colorado
  - Denver Arthritis Clinic, Denver, Colorado
  - Bradenton Research Center, Bradenton, Florida
  - Prohealth Research Center, Doral, Florida
  - LIFE Clinical Trials, Margate, Florida
  - D&H National Research Centers, Miami, Florida
  - IRIS Research and Development, LLC, Plantation, Florida
  - Napa Research Center, Pompano Beach, Florida
  - D&H Tamarac Research Centers, Tamarac, Florida
  - GCP Clinical Research, Tampa, Florida
  - ClinPro Research Solutions, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - MedPharmics, LLC, Metairie, Louisiana
  - MD Medical Research, Oxon Hill, Maryland
  - Santa Fe Rheumatology, Santa Fe, New Mexico
  - Long Island Arthritis & Osteoporosis Care, Babylon, New York
  - Research Carolina Elite, Denver, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Shelby Clinical Research, LLC, Shelby, North Carolina
  - Velocity Clinical Research Cincinnati, Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Chattanooga Research & Medicine PLLC (CHARM), Chattanooga, Tennessee
  - Abigail Rebecca Neiman, MD, PA, Houston, Texas
  - Pioneer Research Solutions Inc - Houston, Houston, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Western Washington Medical Group, Bothell, Washington
  - Arthritis Northwest, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with uncontrolled gout were enrolled at 36 centers across the United States between October 2020 and March 2024.
Pre-assignment Details: A 4-week methotrexate (MTX) run-in period, with a weekly dose of 15 mg, was used to identify screening failures due to MTX intolerance. All participants who completed the run-in period received their first dose of pegloticase on Day 1, followed by additional doses every 2 weeks (Q2W) for a total of 22 weeks.
Groups:
- Pegloticase 60 Minute + MTX: Participants received oral MTX (15 mg) (weekly) during the Run-in Period, then 60-minute pegloticase IV infusions (every 2 weeks) with MTX (weekly) for 24 weeks.
- Pegloticase 45 Minute + MTX: Participants received oral MTX (15 mg) (weekly) during the Run-in Period, then 45-minute pegloticase IV infusions (every 2 weeks) with MTX (weekly) for 24 weeks.
- Pegloticase 30 Minute + MTX: Participants received oral MTX (15 mg) (weekly) during the Run-in Period, then 30-minute pegloticase IV infusions (every 2 weeks) with MTX (weekly) for 24 weeks.
Period: Overall Study
Arm/Group | Pegloticase 60 Minute + MTX | Pegloticase 45 Minute + MTX | Pegloticase 30 Minute + MTX
Started | 116 | 13 | 62
Completed | 96 | 12 | 50
Not Completed | 20 | 1 | 12
Not completed — Lost to Follow-up | 3 | 0 | 4
Not completed — Withdrawal by Subject | 17 | 1 | 8

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) Analysis Set: All participants who received at least 1 dose of pegloticase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegloticase 60 Minute + MTX | Pegloticase 45 Minute + MTX | Pegloticase 30 Minute + MTX | Total
Number analyzed (Participants) | 116 | 13 | 62 | 191
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (11.33) | 61.1 (9.96) | 56.9 (11.04) | 56.2 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 9 | 23
  Male | 104 | 11 | 53 | 168
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 8 | 1 | 2 | 11
  Black or African American | 18 | 3 | 9 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  White | 84 | 9 | 48 | 141
  More than 1 race | 3 | 0 | 1 | 4
  Other | 3 | 0 | 0 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 29 | 1 | 4 | 34
  Not Hispanic or Latino | 87 | 12 | 58 | 157

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced an Infusion Reaction (IR), Including Anaphylaxis, Related to Pegloticase From Day 1 to Week 24
Description: IRs, including anaphylaxis, were assessed after each infusion for a period of 24 weeks. IRs were defined as any infusion-related adverse event (AE) or cluster of temporally-related AEs, not attributable to another cause, which occurred during the pegloticase infusion and up to 2 hours post-infusion. Additional AEs occurring outside of the 2-hour window following infusion could also be categorized as an IR at the Principal Investigator's discretion.
Time Frame: Day 1 to Week 24
Population: Safety Analysis Set (SAS): All participants who received at least 1 dose of pegloticase.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pegloticase 60 Minute + MTX | Pegloticase 45 Minute + MTX | Pegloticase 30 Minute + MTX
Number analyzed (Participants) | 116 | 13 | 62
Percentage of Participants | 6.0 [2.5 to 12.0] | 0 [0.0 to 24.7] | 12.9 [5.7 to 23.9]

2. Secondary Outcome: Percentage of Serum Uric Acid (sUA) Responders at Month 6
Description: Responders were defined as participants who achieved and maintained sUA levels below 6 mg/dL for at least 80% of the time during month 6.
  Responders who met sUA discontinuation criteria (2 consecutive sUA > 6 mg/dL), regardless of treatment status were considered non-responders.
Time Frame: Up to 6 months
Population: mITT Analysis Set: All participants who received at least 1 dose of pegloticase.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pegloticase 60 Minute + MTX | Pegloticase 45 Minute + MTX | Pegloticase 30 Minute + MTX
Number analyzed (Participants) | 116 | 13 | 62
Percentage of Participants | 67.2 [57.9 to 75.7] | 76.9 [46.2 to 95.0] | 56.5 [43.3 to 69.0]

3. Secondary Outcome: Percentage of Participants Who Experienced an IR Leading to Discontinuation of Treatment, Anaphylaxis or Met sUA Discontinuation Criteria
Description: IRs were defined as any infusion-related AE or cluster of temporally-related AEs, not attributable to another cause, which occurred during the pegloticase infusion and for 2 hours post-infusion. Other AEs that occurred outside of the 2 hour window following the infusion may have also been categorized as an IR at the Principal Investigator's discretion.
  Anaphylaxis was defined using the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network criteria.
  Meeting individual sUA discontinuation criteria was defined as two consecutive pre-infusion sUAs > 6 mg/dL after Day 1.
Time Frame: Day 1 to Week 24
Population: SAS: All participants who received at least 1 dose of pegloticase.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pegloticase 60 Minute + MTX | Pegloticase 45 Minute + MTX | Pegloticase 30 Minute + MTX
Number analyzed (Participants) | 116 | 13 | 62
Percentage of Participants | 19.0 [12.3 to 27.3] | 7.7 [0.2 to 36.0] | 32.3 [20.9 to 45.3]

4. Secondary Outcome: Time to First Event of IR Leading to Discontinuation of Treatment, Anaphylaxis or Meeting sUA Discontinuation Criteria in All Participants
Description: Infusion reactions were defined as any infusion-related adverse event or cluster of temporally-related adverse events, not attributable to another cause, which occurred during the infusion and for 2 hours post-infusion. Other adverse events that occurred outside of the 2-hour window following the infusion may have also been categorized as an infusion reaction at the Principal Investigator's discretion.
  Anaphylaxis was defined using the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network criteria.
  Meeting individual serum uric acid discontinuation criteria was defined as two consecutive pre-infusion serum uric acid levels greater than 6 mg/dL after Day 1.
  Time to event was derived as the date of the event minus the date of the first dose of the treatment plus 1. All participants were censored at the date of their last infusion.
Time Frame: Day 1 to Week 24
Population: SAS: All participants who received at least 1 dose of pegloticase.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Pegloticase 60 Minute + MTX | Pegloticase 45 Minute + MTX | Pegloticase 30 Minute + MTX
Number analyzed (Participants) | 116 | 13 | 62
Days | NA [NA to NA] — The median time (95% CI) to occurrence of this composite event was not estimable using Kaplan-Meier analysis due to the low number of these events. | NA [NA to NA] — The median time (95% CI) to occurrence of this composite event was not estimable using Kaplan-Meier analysis due to the low number of these events. | NA [NA to NA] — The median time (95% CI) to occurrence of this composite event was not estimable using Kaplan-Meier analysis due to the low number of these events.

5. Secondary Outcome: Time to First Event of IR Leading to Discontinuation of Treatment, Anaphylaxis or Meeting sUA Discontinuation Criteria in Participants With an Event
Description: IRs were defined as any infusion-related adverse event or cluster of temporally-related adverse events, not attributable to another cause, which occurred during the infusion and for 2 hours post-infusion. Other adverse events that occurred outside of the 2-hour window following the infusion may have also been categorized as an infusion reaction at the Principal Investigator's discretion.
  Anaphylaxis was defined using the National Institute of Allergy and Infectious Diseases/Food Allergy and Anaphylaxis Network criteria.
  Meeting individual serum uric acid discontinuation criteria was defined as two consecutive pre-infusion serum uric acid levels greater than 6 mg/dL after Day 1.
  Time to event was derived as the date of the event minus the date of the first dose of the treatment plus 1. Only participants who experienced an event were included in this analysis.
Time Frame: Day 1 to Week 24
Population: All participants who received at least 1 dose of pegloticase and experienced an IR leading to discontinuation of treatment, anaphylaxis or met sUA discontinuation criteria.
Measure: Median (Full Range); unit: Days
Arm/Group | Pegloticase 60 Minute + MTX | Pegloticase 45 Minute + MTX | Pegloticase 30 Minute + MTX
Number analyzed (Participants) | 22 | 1 | 20
Days | 17.0 [1 to 113] | 15.0 [15 to 15] | 43.0 [15 to 144]

ADVERSE EVENTS:
Time Frame: Up to approximately 1 year.
Description: A 4-week MTX run-in period (15 mg weekly) was conducted to identify screening failures due to MTX intolerance. Of 215 participants receiving MTX, 24 discontinued before receiving pegloticase and were deemed screen failures. The remaining 191 participants completed the run-in period, received pegloticase on Day 1, and were considered enrolled in the trial. All enrolled participants received the first pegloticase dose on Day 1, followed by additional doses Q2W for a total of 22 weeks.
Groups:
- MTX Run-In: MTX Run-In Period
Arm/Group | MTX Run-In | Pegloticase 60 Minute + MTX | Pegloticase 45 Minute + MTX | Pegloticase 30 Minute + MTX
All-Cause Mortality (participants affected / at risk) | 0/215 | 0/116 | 0/13 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/215 | 4/116 | 0/13 | 5/62
Other Adverse Events (participants affected / at risk) | 79/215 | 86/116 | 13/13 | 46/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MTX Run-In (N=215) | Pegloticase 60 Minute + MTX (N=116) | Pegloticase 45 Minute + MTX (N=13) | Pegloticase 30 Minute + MTX (N=62)
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Shigella infection (Infections and infestations) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MTX Run-In (N=215) | Pegloticase 60 Minute + MTX (N=116) | Pegloticase 45 Minute + MTX (N=13) | Pegloticase 30 Minute + MTX (N=62)
Lacrimation increased (Eye disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2 | 4
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 2 | 4 | 0 | 6
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 6 | 0 | 7
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 1 | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 72 | 77 | 9 | 44
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT04511702/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT04511702/SAP_001.pdf